CLINICAL TRIAL: NCT03514420
Title: An Open-label Phase 2 Study of ISIS 703802 (AKCEA-ANGPTL3-LRx) Administered Subcutaneously to Subjects With Familial Partial Lipodystrophy
Brief Title: Study of AKCEA-ANGPTL3-LRx (ISIS 703802) in Participants With Familial Partial Lipodystrophy (FPL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 703802-CS5
Record Dates: First submitted 2018-04-21; First posted 2018-05-02 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Familial Partial Lipodystrophy
Keywords: Lipodystrophy; Lipodystrophy, Familial Partial; Lipid Metabolism Disorders; Dyslipidemias; Kobberling-Dunnigan syndrome (type 1 and 2); Lipoatrophic Diabetes
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Lipodystrophy; Lipid Metabolism Disorders; Dyslipidemias; Diabetes Mellitus, Lipoatrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AKCEA-ANGPTL3-LRx 20 mg (Experimental): Participants received AKCEA-ANGPTL3-LRx 20 milligrams (mg) administered every week for 26 weeks by subcutaneous (SC) injection.
  Interventions: Drug: AKCEA-ANGPTL3-LRx

INTERVENTIONS:
Drug: AKCEA-ANGPTL3-LRx — AKCEA-ANGPTL3-LRx solution for SC injection.
  Other Names: ISIS 703802

SUMMARY:
This is a single-center, open-label study to evaluate the efficacy of AKCEA-ANGPTL3-LRx for reduction of fasting triglycerides in participants with familial partial lipodystrophy.

ELIGIBILITY:
Key Inclusion Criteria:

* Must give written informed consent to participate in the study.
* Clinical diagnosis of familial partial lipodystrophy plus diagnosis of type 2 diabetes mellitus and hypertriglyceridemia.
* Diagnosis of diabetes mellitus, made at least 6 months prior to the Screening with hemoglobin A1c (HbA1c) ≥ 7% to ≤ 12% at Screening and on anti-diabetic therapy as defined in study protocol.
* Hypertriglyceridemia as defined by fasting triglycerides (TG) levels ≥ 500 milligrams per deciliter (mg/dL) at both Screening and Qualification visits. Participants with the clinical diagnosis of FPL and with fasting TG levels ≥ 200 (≥ 2.26 millimoles per liter [mmol/L]) to < 500 mg/dL (≥ 5.7 mmol/L) who meet the genetic or family history criteria for study inclusion may be further screened and enrolled in the study.
* Presence of hepatosteatosis (fatty liver), as evidenced by a Screening magnetic resonance imaging (MRI) indicating a hepatic fat fraction (HFF) ≥ 6.4%.

Key Exclusion Criteria:

* Diagnosis of generalized lipodystrophy.
* Diagnosis of acquired partial lipodystrophy (APL).
* Acute pancreatitis within 4 weeks of Screening.
* Acute coronary syndrome within 6 months of Screening.
* Major surgery within 3 months of Screening.
* Have any other conditions in the opinion of the investigator which could interfere with the participant participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States of America from 15 June 2018 to 21 August 2019.
Pre-assignment Details: A total of 8 participants diagnosed with familial partial lipodystrophy (FPL) were screened, out of which 4 participants were treated with AKCEA-ANGPTL3-LRx 20 milligrams (mg). All 4 participants completed the study.
Groups:
- AKCEA-ANGPTL3-LRx 20 mg: Participants received AKCEA-ANGPTL3-LRx 20 mg administered every week for 26 weeks by subcutaneous (SC) injection.
Period: Overall Study
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- AKCEA-ANGPTL3-LRx 20 mg: Participants received AKCEA-ANGPTL3-LRx 20 mg administered every week for 26 weeks by SC injection.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (3.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] | 817.8 (431.89)
Fasting Apolipoprotein B-48 (Apo B-48) [Mean (Standard Deviation); unit: mg/dL] | 5.109 (0.5588)
Fasting Apolipoprotein C-III (Apo CIII) [Mean (Standard Deviation); unit: mg/dL] | 28.435 (11.8481)
Fasting Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 124.95 (24.972)
Fasting Non-High Density Lipoprotein- Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 223.4 (22.03)
Fasting High Density Lipoprotein- Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 25.13 (3.473)
Fasting Apolipoprotein A-I (Apo A-1) [Mean (Standard Deviation); unit: mg/dL] | 121.3 (9.67)
Fasting Very low Density Lipoprotein-Cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] — VLDL-C calculated using direct test method. Population: Number analyzed signifies the number of participants with data available for fasting VLDL-C.
  mg/dL
    number analyzed (Participants) | 3
    (all) | 130.3 (22.90)
Fasting Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — LDL-C calculated using ultracentrifugation method. Population: Number analyzed signifies the number of participants with data available for fasting LDL-C.
  mg/dL
    number analyzed (Participants) | 3
    (all) | 93.3 (24.38)
Area Under Curve (AUC) of Plasma Glucose [Mean (Standard Deviation); unit: milligram/deciliter*minute (mg/dL*min)] | 257 (45.2622)
AUC of Serum Insulin [Mean (Standard Deviation); unit: milli international units/ liter*minute] | 42.625 (4.852748)
AUC of Serum C-peptide [Mean (Standard Deviation); unit: nanogram/milliliter*minute (ng/mL*min)] — Population: Number analyzed signifies the number of participants with data available for AUC of Serum C-peptide.
  nanogram/milliliter*minute (ng/mL*min)
    number analyzed (Participants) | 3
    (all) | 3.266 (1.234)
AUC of Free Fatty Acid [Mean (Standard Deviation); unit: milliequivalents/liter*min (mEq/L*min)] — Population: Number analyzed signifies the number of participants with data available for AUC of Free fatty acid.
  milliequivalents/liter*min (mEq/L*min)
    number analyzed (Participants) | 3
    (all) | 1.57 (0.458)
AUC of Gastric Inhibitory Polypeptide (GIP) [Mean (Standard Deviation); unit: picograms/milliliter*minute (pg/mL*min)] — Population: Number analyzed signifies the number of participants with data available for AUC of GIP.
  picograms/milliliter*minute (pg/mL*min)
    number analyzed (Participants) | 3
    (all) | 46.02 (38.555)
AUC of Glucagon-like Peptide 1 (GLP-1) [Mean (Standard Deviation); unit: picomoles/liter*minute (pmol/L*min)] — Population: Number analyzed signifies the number of participants with data available for AUC of GLP-1.
  picomoles/liter*minute (pmol/L*min)
    number analyzed (Participants) | 3
    (all) | 23.35 (17.065)
AUC of Peptide Tyrosine Tyrosine (PYY) [Mean (Standard Deviation); unit: pg/mL*min] | 80.412 (99.559)
AUC of Serum Ghrelin [Mean (Standard Deviation); unit: pg/mL*min] | 27.955 (15.127)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Triglycerides Levels at End of the Treatment (Week 27)
Description: The baseline was defined as the average of Day 1 pre-dose fasting assessment and the last fasting measurement prior to Day 1 pre-dose fasting assessment.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
percent change | -59.9 (26.29)

2. Secondary Outcome: Change From Baseline in Area Under the Curve (AUC) of Plasma Glucose as Assessed by Mixed Meal Test (MMT) at End of the Treatment
Description: Change from Baseline to Week 27 in the area under the curve (AUC) of Plasma Glucose was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
mg/dL*min | -9815.0 (4071.43)

3. Secondary Outcome: Change From Baseline in AUC of Serum Insulin as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of Serum Insulin was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milli international units per liter*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
milli international units per liter*min | 3262.0 (3775.09)

4. Secondary Outcome: Change From Baseline in AUC of Serum C-peptide as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of Serum C-peptide was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
ng/mL*min | -192.3 (257.10)

5. Secondary Outcome: Change From Baseline in AUC of Free Fatty Acid (FFA) as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of FFA was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mEq/L*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
mEq/L*min | -60.0 (42.52)

6. Secondary Outcome: Change From Baseline in AUC of Serum Ghrelin as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of Serum Ghrelin was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
pg/mL*min | 8479.5 (7241.20)

7. Secondary Outcome: Change From Baseline in AUC of Incretin Hormone (Gastric Inhibitory Polypeptide [GIP]) as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of Incretin Hormone: GIP was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 2
pg/mL*min | -1694.7 (11752.50)

8. Secondary Outcome: Change From Baseline in AUC of Incretin Hormone (Glucagon-like Peptide -1 [GLP-1]) as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of Incretin Hormone: GLP-1 was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
pmol/L*min | 1677.3 (11301.79)

9. Secondary Outcome: Change From Baseline in AUC of Peptide Tyrosine Tyrosine (PYY) as Assessed by MMT at End of the Treatment
Description: Change from Baseline to Week 27 in the AUC of PYY was assessed.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL*min
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
pg/mL*min | 6549.0 (10632.50)

10. Secondary Outcome: Change From Baseline in HDL-C at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | 2.1 (6.88)

11. Secondary Outcome: Change From Baseline in LDL-C at End of the Treatment
Description: The baseline was defined as the average of Day 1 pre-dose fasting assessment and the last fasting measurement prior to Day 1 pre-dose fasting assessment. LDL-C calculated using ultracentrifugation method.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 1
mg/dL | 24.0 (NA) — Due to a single analyzed participant, standard deviation was not calculated.

12. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -42.3 (32.29)

13. Secondary Outcome: Change From Baseline in VLDL-C at End of the Treatment
Description: The baseline was defined as the average of Day 1 pre-dose fasting assessment and the last fasting measurement prior to Day 1 pre-dose fasting assessment. VLDL-C was calculated using direct test method.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 1
mg/dL | -32.0 (NA) — Due to a single analyzed participant, standard deviation was not calculated.

14. Secondary Outcome: Change From Baseline in Non-HDL-C at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -44.4 (34.27)

15. Secondary Outcome: Change From Baseline in ApoB at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | 1.25 (25.265)

16. Secondary Outcome: Change From Baseline in ApoB-48 at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -3.601 (1.3284)

17. Secondary Outcome: Change From Baseline in Apolipoprotein B 100 (ApoB-100) at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | 4.433 (24.6001)

18. Secondary Outcome: Change From Baseline in ApoA-1 at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -20.8 (22.92)

19. Secondary Outcome: Change From Baseline in ApoC-III at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -13.555 (9.1220)

20. Secondary Outcome: Change From Baseline in ApoC-III: Chylomicron at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Data is not available as the collected Baseline samples were not sufficient to assess this outcome measure.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

21. Secondary Outcome: Change From Baseline in ApoC-III: VLDL at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Data is not available as the collected Baseline samples were not sufficient to assess this outcome measure.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

22. Secondary Outcome: Change From Baseline in ApoC-III: LDL at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 1
mg/dL | -2.110 (NA) — Due to a single analyzed participant, standard deviation was not calculated.

23. Secondary Outcome: Change From Baseline in ApoC-III: HDL at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
mg/dL | -9.904 (5.9174)

24. Secondary Outcome: Change From Baseline in Lipoprotein a (Lp[a]) at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
nanomoles per liter (nmol/L) | 8.4 (14.99)

25. Secondary Outcome: Change From Baseline in Free Fatty Acid (FFA) at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
millimoles per liter (mmol/L) | -0.5779 (0.8778)

26. Secondary Outcome: Change From Baseline in Glycerol Levels at End of the Treatment
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromoles per liter (μmol/L)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
micromoles per liter (μmol/L) | -8.0 (3.32)

27. Secondary Outcome: Change From Baseline in Lipoprotein Particle Size at End of the Treatment
Description: The baseline was defined as the Day 1 pre-dose fasting assessment. Lipoprotein Particle size included: HDL size, LDL size and VLDL size.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nanometer (nm)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
nanometer (nm)
  HDL Size | 0.1 (0.44)
  LDL Size | 0.2 (0.48)
  VLDL Size | -8.7 (7.63)

28. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at End of the Treatment
Description: The baseline was defined as the last non-missing assessment prior to the first dose of study drug.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
percentage of HbA1c | -0.23 (0.991)

29. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment-Estimated Insulin Resistance (HOMA-IR)
Description: as for outcome 1
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Due to the low number of participants, data for this outcome measure was not collected.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

30. Secondary Outcome: Change From Baseline in Adiponectin at End of the Treatment
Description: The baseline was defined as the Day 1 pre-dose fasting assessment.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
microgram per milliliter (µg/mL) | 0.08 (0.742)

31. Secondary Outcome: Change From Baseline in and Leptin at End of the Treatment
Description: The baseline was defined as the Day 1 pre-dose fasting assessment
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
nanogram per milliliter (ng/mL) | -0.19 (2.650)

32. Secondary Outcome: Change From Baseline in Hepatic Fat Fraction (HFF) as Assessed by Magnetic Resonance Imaging (MRI) at End of the Treatment
Description: The baseline was defined as the last non-missing assessment prior to the first dose of study drug.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
percentage of hepatic fat | -1.1400 (6.1107)

33. Secondary Outcome: Changes From Baseline in Body Fat Distribution for Various Areas in the Body as Measured by Skinfold Thickness at End of the Treatment
Description: The baseline was defined as the last assessment prior to the first dose of study drug. Change in body fat distribution was measured as right anterior thigh skinfold thickness and right tricep skinfold thickness by Skinfold Thickness.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
millimeter (mm)
  Right Anterior Thigh Skinfold Thickness | 1.6 (2.38)
  Right Tricep Skinfold Thickness | -2.1 (3.76)

34. Secondary Outcome: Changes From Baseline in Body Fat Distribution for Various Areas in the Body as Measured by Dual-Energy X-ray Absorptiometry (DEXA) at End of the Treatment
Description: The baseline was defined as the Screening assessment. Change in body fat distribution (arm bone mass, arm fat mass, arm lean mass, arm total mass, leg bone mass, leg fat mass, leg lean mass, leg total mass, total bone mass, total fat mass, total lean mass, total total mass , trunk bone mass, trunk fat mass, trunk lean mass and trunk total mass) was measures obtained from DEXA.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
gram (g)
  Arm Bone Mass | 11.3 (19.86)
  Arm Fat Mass | 603.8 (803.36)
  Arm Lean Mass | 273.3 (612.04)
  Arm Total Mass | 875.0 (1384.14)
  Leg Bone Mass | 16.5 (40.53)
  Leg Fat Mass | 436.8 (662.80)
  Leg Lean Mass | -345.8 (1384.52)
  Leg Total Mass | 125.0 (1736.62)
  Total Bone Mass | 37.3 (77.03)
  Total Fat Mass | 1197.3 (1667.27)
  Total Lean Mass | -891.5 (1852.25)
  Total Total Mass | 350.0 (3183.81)
  Trunk Bone Mass | 23.3 (35.37)
  Trunk Fat Mass | 183.5 (296.49)
  Trunk Lean Mass | -728.8 (590.17)
  Trunk Total Mass | -500.0 (836.66)

35. Secondary Outcome: Changes From Baseline in Body Fat Distribution for Total Bone Mineral Density in the Body as Measured by Dual-Energy X-ray Absorptiometry (DEXA) at End of the Treatment
Description: The baseline was defined as Screening assessment. Change in body fat distribution for total Bone mineral density was measures obtained from DEXA.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: gram per centimeter square (g/cm^2)
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
gram per centimeter square (g/cm^2) | 0.0 (0.07)

36. Secondary Outcome: Change From Baseline in Visceral Adipose Tissue (VAT) as Measured by Magnetic Resonance Imaging (MRI) at End of the Treatment
Description: The baseline was defined as the last assessment prior to the first dose of study drug.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Due to the low number of participants, data for this outcome measure was not collected.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

37. Secondary Outcome: Change From Baseline in Subcutaneous Adipose Tissue (SAT) as MRI at End of the Treatment
Description: The baseline was defined as the last assessment prior to the first dose of study drug.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Due to the low number of participants, data for this outcome measure was not collected.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

38. Secondary Outcome: Change From Baseline in Body Weight at End of the Treatment
Description: The baseline was defined as the Day 1 pre-dose assessment.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
kg | -1.05 (3.309)

39. Secondary Outcome: Change From Baseline in Waist Circumference at End of the Treatment
Description: The baseline was defined as the Screening assessment.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
cm | -1.88 (1.863)

40. Secondary Outcome: Change From Baseline in Waist/Hip Ratio at End of the Treatment
Description: The baseline was defined as screening assessment.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Due to the low number of participants, data for this outcome measure was not collected.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 0

41. Secondary Outcome: Change From Baseline in Quality of Life (QoL)
Description: The baseline was defined as the screening assessment. Quality of life measures the severity of fatigue, severity of trouble thinking or remembering and severity of waking up tired in participants, on a scale ranging from 0 to 3, where, 0= No problem, 1= Mild, 2= Moderate and 3= severe. Higher scores indicates more severity or more impact on quality of life.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
Participants
  Severity of fatigue: Improved | 1
  Severity of fatigue: Worse | 1
  Severity of fatigue: No change | 2
  Severity of trouble thinking or remembering: Improved | 0
  Severity of trouble thinking or remembering: Worse | 0
  Severity of trouble thinking or remembering: No change | 4
  Severity of waking up tired: Improved | 1
  Severity of waking up tired: Worse | 2
  Severity of waking up tired: No change | 1

42. Secondary Outcome: Change From Baseline in Pain Score at End of the Treatment
Description: The baseline was defined as a Screening assessment. Pain score is used to determine disease activity in participants, on a scale ranging from 0 to 5 where 0= never, 1= hardly noticed, 2= slightly, 3= moderately, 4= strongly, and 5= very strongly where higher scores indicated higher degree of pain.
Time Frame: Baseline and End of the Treatment (Week 27)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
score on a scale | -3.8 (3.50)

43. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. "A treatment-emergent adverse event (TEAE) is defined as any AE starting on or after the first dose of the study drug
Time Frame: From signing of informed consent to end of follow up period (Up to week 40)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: From signing of informed consent to end of follow up period (Up to week 40)
Description: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKCEA-ANGPTL3-LRx 20 mg (N=4)
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Troponin increased (Investigations) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AKCEA-ANGPTL3-LRx 20 mg (N=4)
Hot flush (Vascular disorders) | 1
Albumin urine present (Investigations) | 3
Antinuclear antibody positive (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Hepatic steatosis (Hepatobiliary disorders) | 2
Blood magnesium decreased (Investigations) | 3
Creatinine urine increased (Investigations) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Fatigue (General disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
International normalised ratio increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Oedema peripheral (General disorders) | 1
Insulin C-peptide decreased (Investigations) | 1
Urine albumin/creatinine ratio increased (Investigations) | 2
Depression (Psychiatric disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
urinary casts (Investigations) | 2
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Blood creatinine increased (Investigations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Mean cell haemoglobin decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Mean cell volume decreased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Injection site dryness (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Crystal urine present (Investigations) | 1
Liver function test (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03514420/Prot_SAP_000.pdf